CLINICAL TRIAL: NCT05332509
Title: Mobility and Quality of Life in Community Ambulators With Knee Locking Deficiency Using a Microprocessor Controlled Knee Ankle Foot Orthosis and a Stance Control Orthosis: Randomized Crossover Trial
Brief Title: C-BRACE Versus SCO in Community Ambulators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock France SNC (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BP-11-PT007; 2022-A00116-37 (Other: ANSM)
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Lower Limb; Pareses
Keywords: Knee-ankle-foot orthosis; KAFO
MeSH Terms: conditions — Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-BRACE/SCO (Experimental): The patient is first fitted during 2 months with the C-BRACE orthosis, them, after 2 weeks wash-out period, the patient is fitted with its Stance Controlled Orthosis (SCO).
  Interventions: Device: C-BRACE; Device: SCO
- SCO/C-BRACE (Other): The patient is using its Stance controlled orthosis (SCO) during 2 months, then, after 2 weeks wash-out period, the patient is fitted with the C-BRACE orthosis.
  Interventions: Device: C-BRACE; Device: SCO

INTERVENTIONS:
Device: C-BRACE — The C-BRACE is a custom made Knee-Ankle-Foot-Orthosis with a microprocessor-controlled hydraulic knee-joint articulation. The C-BRACE technology offers to a patient with knee locking deficiencies the following advantages: approximation of the physiological gait pattern, stability while standing and walking, adaptation to various surfaces, inclines, gait situations and walking speeds.
Device: SCO — The SCO is a custom made Knee-Ankle-Foot-Orthosis with a knee-joint locked during stance phase and released during swing phase.

SUMMARY:
The purpose of this multicentric study is to assess the impact of C-BRACE on mobility, endurance, confidence, participation, satisfaction, psychosocial adjustment and quality of life in community ambulators using a Stance Control Orthosis.

DETAILED DESCRIPTION:
During two months of inclusion period, the investigators invite all patients matching with inclusion criteria for an enrolment visit, collect written consent and record general patient information. The eCRF (electronic Case Report Form) assigns the enrolled patient into one group for the trial (C-BRACE/SCO or SCO/C-BRACE), in a randomized order. The assessments are performed after 2 month follow-up period with each orthosis with a minimal wash-out period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* person with knee locking deficiency
* person using a SCO (Stance Control Orthosis) for at least three months, walking with a swing phase on a flat ground, without walking aid or with one cane or one crutch.
* person having the ability to walk at 3km/h (measured with 10 meters walk test) with the SCO in unlocked mode.
* person with a stable stance phase on the contralateral side

Exclusion Criteria:

* person with deficient or unstable contralateral knee, including person using a Knee-Ankle Foot Orthosis on the contralateral limb
* person walking using two canes, two crutches, one or two underarm crutches or a walker
* person with health condition not compatible with the study protocol
* person under 18 years old
* person unwilling / unable to follow the entire study protocol / instructions
* person who did not give her written consent to participate to the study or unable to personally give her consent
* person with knee and/or hip flexion contracture >10°
* person with genu varum / valgum > 10° (not reducible)
* person with moderate to severe spasticity
* person with leg length discrepancy > 15cm
* person who necessitate the use of an orthoprosthesis
* person with body weight > 125kg
* person with unstable trunk in standing position
* person with cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
PLUS-M™ - Mobility | 2-months
  12-items Self-reported measure of mobility as the ability to move intentionally and independently from one place to another.

SECONDARY OUTCOMES:
6 minutes walk test | 2-months
  Distance walked in 6 minutes
ABC-s Activities-specific Balance Confidence - simplified | 2-months
  15-items self-reported measure of the perceived balance confidence an individual has while completing various ambulatory activities on 4-levels scale.
PSFS - Patient Specific Functional Scale | 2-months
  Patients will be asked to identify three activities that they are having difficulty or are unable to perform because of their condition. Patients will then be asked to rate their ability to perform each activity on a numerical scale ('0' being unable to perform the activity, and '10' being able to full perform the activity).
PIADS - Psychosocial Impact of Assistive Devices Scale | 2-months
  26-items questionnaire that assess the effects of an assistive device on functional independence, well-being and quality of life from the person's disability's point of view. Each item is noted on a 7-points Likert scale going from -3 (maximum negative impact) to +3 (maximum positive impact).
EQ-5D-5L - Quality of Life | 2-months
  Self-reported measure of health status composed of 5 dimensions: mobility, ability to self-care, ability to undertake usual activities, pain and discomfort, anxiety and depression. Each dimension is rated on a 5-point scale.
QUEST 2.0 - Satisfaction | 2-months
  12-items self-reported measure on patient's satisfaction regarding the technology of the device and the services around the device. It allows the patient to express himself on the 3 most important criteria to him.

CONTACTS AND LOCATIONS:
Overall Officials: François GENET, Prof. med, Study Chair — CHU Raymond Poincaré Garches France; Frank BRAATZ, Prof. med, Study Chair — PFH Private Hochschule Göttingen Germany; Axel RUETZ, Dr. med., Study Chair — Katholisches Klinikum Koblenz-Montabaur Germany
Locations (18):
- France (16):
  - CRF Korian Le Mont Veyrier, Argonay
  - Centre Jacques Calvé Fondation Hopale, Berck
  - HIA Percy, Clamart
  - Pôle de Réadaptation de Cornouaille, Concarneau
  - Centre Hospitalier Dieppe, Dieppe
  - Hôpital Raymond-Poincaré, Garches
  - Hia Laveran, Marseille
  - IRR Louis Pierquin, Nancy
  - CRRF La Chataigneraie, Paris
  - CRRF Léopold Bellan, Paris
  - Centre Bouffard Vercelli, Perpignan
  - CRRF La Tourmaline, Saint-Herblain
  - CRF Salies de Béarn, Salies-de-Béarn
  - LADAPT Thionis, Thionville
  - Chu Rangueil, Toulouse
  - IRMA Institut Robert Merle d'Aubigné, Valenton
- Germany (2):
  - PFH Private Hochschule Göttingen, Göttingen
  - Katholisches Klinikum Koblenz-Montabaur, Koblenz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deems-Dluhy S, Hoppe-Ludwig S, Mummidisetty CK, Semik P, Heinemann AW, Jayaraman A. Microprocessor Controlled Knee Ankle Foot Orthosis (KAFO) vs Stance Control vs Locked KAFO: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Feb;102(2):233-244. doi: 10.1016/j.apmr.2020.08.013. Epub 2020 Sep 22. PMID 32976844
- [Background] Karatzios C, Loiret I, Luthi F, Leger B, Le Carre J, Saubade M, Muff G, Benaim C. Transcultural adaptation and validation of a French version of the Prosthetic Limb Users Survey of Mobility 12-item Short-Form (PLUS-M/FC-12) in active amputees. Ann Phys Rehabil Med. 2019 May;62(3):142-148. doi: 10.1016/j.rehab.2019.02.006. Epub 2019 Apr 6. PMID 30965157
- [Background] Chatman AB, Hyams SP, Neel JM, Binkley JM, Stratford PW, Schomberg A, Stabler M. The Patient-Specific Functional Scale: measurement properties in patients with knee dysfunction. Phys Ther. 1997 Aug;77(8):820-9. doi: 10.1093/ptj/77.8.820. PMID 9256870
- [Background] Demers L, Monette M, Descent M, Jutai J, Wolfson C. The Psychosocial Impact of Assistive Devices Scale (PIADS): translation and preliminary psychometric evaluation of a Canadian-French version. Qual Life Res. 2002 Sep;11(6):583-92. doi: 10.1023/a:1016397412708. PMID 12206579
- [Background] Middleton A, Fritz SL, Lusardi M. Walking speed: the functional vital sign. J Aging Phys Act. 2015 Apr;23(2):314-22. doi: 10.1123/japa.2013-0236. Epub 2014 May 2. PMID 24812254
- [Background] Probsting E, Kannenberg A, Zacharias B. Safety and walking ability of KAFO users with the C-Brace(R) Orthotronic Mobility System, a new microprocessor stance and swing control orthosis. Prosthet Orthot Int. 2017 Feb;41(1):65-77. doi: 10.1177/0309364616637954. Epub 2016 Jul 10. PMID 27151648
- [Background] Schmalz T, Probsting E, Auberger R, Siewert G. A functional comparison of conventional knee-ankle-foot orthoses and a microprocessor-controlled leg orthosis system based on biomechanical parameters. Prosthet Orthot Int. 2016 Apr;40(2):277-86. doi: 10.1177/0309364614546524. Epub 2014 Sep 23. PMID 25249381
- [Background] Filiatrault J, Gauvin L, Fournier M, Parisien M, Robitaille Y, Laforest S, Corriveau H, Richard L. Evidence of the psychometric qualities of a simplified version of the Activities-specific Balance Confidence scale for community-dwelling seniors. Arch Phys Med Rehabil. 2007 May;88(5):664-72. doi: 10.1016/j.apmr.2007.02.003. PMID 17466738
- [Background] Andrade LF, Ludwig K, Goni JMR, Oppe M, de Pouvourville G. A French Value Set for the EQ-5D-5L. Pharmacoeconomics. 2020 Apr;38(4):413-425. doi: 10.1007/s40273-019-00876-4. PMID 31912325